CLINICAL TRIAL: NCT05160142
Title: Diabetes Inspired Culinary Education
Acronym: DICE
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Responsible Party: Principal Investigator, Catherine Rogers, Assistant Professor, Case Western Reserve University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY20190718
Record Dates: First submitted 2019-05-17; First posted 2021-12-16 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Type I Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Single group pretest-poshest study design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Participate in the DICE program, which entails culinary and diabetes educational programming delivered weekly for 10 consecutive weeks.
  Interventions: Behavioral: DICE

INTERVENTIONS:
Behavioral: DICE — 10-week culinary and nutrition education program for children with type I diabetes

SUMMARY:
The aim of this study is to assess the feasibility and efficacy of a community-based culinary nutrition education program (Diabetes Inspired Culinary Education, DICE) on improving the diabetes management and dietary intake of 6-14 year old children with type I diabetes mellitus (TIDM).

ELIGIBILITY:
Inclusion Criteria:

* Children: 6-14 years old; diagnosed with type I diabetes within the past 5 years; English speaking
* Adults: primary caregiver of a 6-14 year old child diagnosed with type I diabetes within the past 5 years; English speaking

Exclusion Criteria:

-

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-09-05 (Actual); Primary Completion 2019-11-21 (Actual); Study Completion 2019-11-21 (Actual)

PRIMARY OUTCOMES:
% Change in Hemoglobin A1c | Baseline/pretest, 3 months/posttest
  Blood glucose/diabetes management

SECONDARY OUTCOMES:
Change in daily servings of fruit | Baseline/pretest, 3 months/posttest
  Daily fruit intake assessed via 3, 24-hour dietary recalls collected electronically using the Automated Self-Assessment 24-hour (ASA-24) dietary assessment tool
Change in daily servings of vegetables | Baseline/pretest, 3 months/posttest
  Daily vegetable intake assessed via 3, 24-hour dietary recalls collected electronically using the Automated Self-Assessment 24-hour (ASA-24) dietary assessment tool
Change in daily servings of whole grains | Baseline/pretest, 3 months/posttest
  Daily whole grain intake assessed via 3, 24-hour dietary recalls collected electronically using the Automated Self-Assessment 24-hour (ASA-24) dietary assessment tool
Change in daily servings of sugar-sweetened beverages | Baseline/pretest, 3 months/posttest
  Daily sugar-sweetened beverage intake assessed via 3, 24-hour dietary recalls collected electronically using the Automated Self-Assessment 24-hour (ASA-24) dietary assessment tool
Change in daily total caloric intake | Baseline/pretest, 3 months/posttest
  Daily caloric intake assessed via 3, 24-hour dietary recalls collected electronically using the Automated Self-Assessment 24-hour (ASA-24) dietary assessment tool
Change in primary caregiver body mass index (kg/m2) | Baseline/pretest, 3 months/posttest
  Assessment of weight status using calibrated stadiometer and electronic scale.
Change in child body mass index z-score | Baseline/pretest, 3 months/posttest
  Assessment of weight status using calibrated stadiometer and electronic scale.
Change in child blood pressure z-score | Baseline, 3 months, 6 months, 9 months
  Includes systolic and diastolic blood pressure z-scores
Change in child food preparation attitude, self-efficacy and frequency of involvement | Baseline/pretest, 3 months/posttest
  Scale 0-132 (higher score indicates more positive attitude, higher self-efficacy, greater frequency of involvement)
Change in child adherence to TIDM management regimen score | Baseline/pretest, 3 months/posttest
  Assessed via Diabetes Management Questionnaire - Scale of 14-70 (higher score indicating greater adherence to management regimen)
Change in child quality of life score | Baseline/pretest, 3 months/posttest
  Assessed via Diabetes Quality of Life for Youth questionnaire - Scale of 41-205 (higher score indicating better quality of life)
Change in primary caregiver self-efficacy for diabetes management score | Baseline/pretest, 3 months/posttest
  Assessed via Maternal Self-Efficacy for Diabetes Management Scale - Scale of 8-40 (higher score indicating greater self-efficacy for diabetes management)
Change in primary caregiver self-efficacy for healthy meal planning and eating score | Baseline/pretest, 3 months/posttest
  Assessed via Parent Mealtime Self-Efficacy Questionnaire - Scale of 11-55 (higher score indicating greater self-efficacy for healthy meal planning and eating)

CONTACTS AND LOCATIONS:
Locations (1):
- Dave's Grocery Store and Teaching Kitchen, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No